CLINICAL TRIAL: NCT01858155
Title: Phase I Dose Finding Study for Melatonin in Pediatric Oncology Patients With Relapsed Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: C17 Council (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: C17 MEL P1
Record Dates: First submitted 2013-05-15; First posted 2013-05-21 (Estimated); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Relapsed Malignant Solid Tumor
MeSH Terms: interventions — Melatonin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Melatonin (Experimental)
  Interventions: Drug: Melatonin

INTERVENTIONS:
Drug: Melatonin
  Other Names: SISU Melatonin

SUMMARY:
This study will evaluate dose escalation of melatonin in pediatric oncology patients with relapsed solid tumors. The purpose of this study is to determine the safety of melatonin at a dose up to 20 mg daily, as well as to determine the maximum tolerated dose of melatonin.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be able to take medication by mouth either by swallowing, chewing or sublingual routes.
* Patients must have a documented life expectancy of ≥ 8 weeks.
* Patients must have histologic or radiographic evidence of a relapsed malignant solid tumor. Intrinsic brain stem tumors or optic pathway gliomas may be diagnosed by clinical and radiologic methods.
* Patient, parent, legal representative and/or guardian must sign a written informed consent. Assent, when appropriate, will be obtained according to institutional guidelines.
* Minimum Weight Requirements: Dose level 1 - 22.2kg, Dose level 2 - 11.1kg, Dose level 3 - 5.6kg
* Patients must be taking a stable dose (with no additions, modifications or deletions) of chemotherapy started ≥ 14 days prior study enrollment.
* Prescribed Chemotherapy drug(s) must not be known to interact with melatonin
* Adequate Bone Marrow Function Defined as:

  1. Patients with solid tumors without bone marrow involvement:

     * Peripheral absolute neutrophil count (ANC) ≥ 1 x109/L
     * Platelet count ≥ 50 X 109/L (transfusion independent, defined as not receiving platelet transfusions within a 7 day period prior to enrollment)
     * Hemoglobin ≥ 80 g/L (may receive RBC transfusions)
  2. Patients with known bone marrow metastatic disease are eligible for study but not evaluable for hematologic toxicity.

     * Must not be known to be refractory to red cell or platelet transfusions.
     * These patients do not need to meet the bone marrow function requirements, as hematological toxicity will not be measured due to metastatic disease.
* Adequate Liver Function Defined as:

  * Total Bilirubin ≤ 1.5 x upper limit of normal (ULN) for age.
  * ALT ≤ 1.5 x ULN for age.

Exclusion Criteria:

* Chemotherapy: Melatonin inhibits the action of doxorubicin
* Growth factors that support white cell number administered ≤ 7 days prior to enrollment.
* Patients requiring corticosteroids who are not on a stable or decreasing dose of corticosteroid for ≥ 14 days.
* Patients prescribed immunosuppressant therapy that is not specifically utilized for chemotherapy purposes. Patient prescribed: Cyclosporine, Mycophenolate Mofetil HCL, Tacrolimus, Sirolimus and Azathioprine should be excluded
* Patients prescribed anti-coagulation therapy (Warfarin, Low Molecular Weight Heparin (LMWH), or System Heparin Therapy)
* Concomitant medications that are known CYP1A2 inhibitors interact with Melatonin.
* Patients prescribed megace, corticosteroids and periactin started ≤ 14 days prior to study enrollment.
* Patients taking the following medications: benzodiazepines, nifedipine, NSAID's, ASA and/or Beta Blockers
* Patients ≤ 7 days post-operative from any surgical procedure.
* Patients with any signs of active post-operative bleeding.
* Patients with an infection that is not responding to anti-microbial therapy.
* Any condition that would negatively impact effective gut absorption and/or swallowing of study medication.
* Patients in the opinion of the investigator may not be able to comply with study protocol requirements
* Patients already receiving melatonin are excluded from the study.
* Allergies to the medicinal and/or non-medicinal ingredients of melatonin which include: Melatonin, Calcium Salicate, Croscarmellose Sodium, IsoMalt, Magnesium Stearate, Microcrystalline Cellulose.
* As melatonin can cause fatigue, patients taking melatonin should refrain from driving or operating machinery within 5 hours of taking the melatonin.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 9 (Actual)
Dates: Start 2013-05; Primary Completion 2017-12 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated daily dose of melatonin. | 8 Weeks

SECONDARY OUTCOMES:
Number of dose limiting toxicities during 8 weeks of melatonin therapy. | 8 Weeks
Peak plasma concentration (Cmax) and area under the plasma concentration versus time curve (AUC) of Melatonin. | 8 Weeks
The quantity of cytokines will be measured during 8 weeks of melatonin therapy. | 8 Weeks
Change from Baseline in weight after 8 weeks of therapy. | 8 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Donna Johnston, MD, Principal Investigator — Children's Hospital of Eastern Ontario
Locations (5):
- Canada (5):
  - Alberta Children's Hospital, Calgary, Alberta
  - Children's & Women's Health Centre of British Columbia, Vancouver, British Columbia
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - The Hospital for Sick Children, Toronto, Ontario
  - CHU Ste-Justine, Montreal, Quebec